CLINICAL TRIAL: NCT04524234
Title: Cardiac Dysfunction in Critically Ill Patients With COVID-19
Acronym: CARDYCOVID
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jonatan Oras, Associate professor, Sahlgrenska University Hospital
Other Study IDs: CARDY CRIT COVID
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Left Ventricular Dysfunction; Right Ventricular Dysfunction; Pulmonary Hypertension
MeSH Terms: conditions — COVID-19; Ventricular Dysfunction, Left; Ventricular Dysfunction, Right; Hypertension, Pulmonary | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography for assessment of cardiac function

SUMMARY:
Cardiac dysfunction has been reported to be common in patients infected with COVID-19. The aim of this study is to evaluate the clinical importance of cardiac dysfunction in critically ill patients infected with COVID-19.

DETAILED DESCRIPTION:
Cardiac dysfunction has been reported to be common in patients infected with COVID-19. The aim of this study is to evaluate the clinical importance of cardiac dysfunction in critically ill patients with COVID-19. Patients admitted to the intensive care unit, with COVID-19 are examined with echocardiography for assessment of left and right ventricular dysfunction within 72 hours from admission and repeated after four to seven days.

Cardiac dysfunction was defined as having either left ventricular (LV) dysfunction, defined as having an ejection fraction <50% and/or regional hypokinesia, or right ventricular (RV) dysfunction, defined as having a tricuspid annular plane excursion (TAPSE) <17mm or a moderate/severe RV dysfunction assessed visually.

The cardiac biomarkers troponin and NTproBNP and clinical data are recorded at time of each echo. Mortality status is recorded at 30 days.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to the intensive care unit infected with COVID-19

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to participating unit, being infected with COVID-19 are eligible for inclusion
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  All cause death in patients with vs without cardiac dysfunction

SECONDARY OUTCOMES:
Left ventricular dysfunction | Within 72 hours from admission
  Prevalence of left ventricular dysfunction
Right ventricular dysfunction | Within 72 hours from admission
  Prevalence of right ventricular dysfunction
Risk-factors | Within 72 hours from admission
  Clinical variables associated with risk of having cardiac dysfunction
Cardiac biomarkers | Within 72 hours from admission
  Levels of cardiac biomarkers in patients with vs without cardiac dysfunction
Left ventricular dysfunction | During ICU-stay
  Prevalence of left ventricular dysfunction
Right ventricular dysfunction | During ICU-stay
  Prevalence of right ventricular dysfunction
Risk-factors | During ICU-stay
  Clinical variables associated with risk of having cardiac dysfunction
Cardiac biomarkers | During ICU-stay
  Levels of cardiac biomarkers in patients with vs without cardiac dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Oras, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (5):
- Sweden (5):
  - Södersjukhuset, Stockholm, Region Stockholm
  - Sahlgrenska University Hospital/Mölndal, Gothenburg, Västra Götaland County
  - Sahlgrenska University Hospital/Östra, Gothenburg, Västra Götaland County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - North Älvsborg County Hospital, Trollhättan, Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: Undecided